CLINICAL TRIAL: NCT06468449
Title: Effects of Optimal Load Strength Training on Muscle Power Output and Neuromuscular Adaptation During Takeoff Among China University Long Jump Athletes
Brief Title: Strength Training on Muscle Power Output and Neuromuscular Adaptation Among China University Long Jump Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rong Wenchao (Other)
Responsible Party: Sponsor-Investigator, Rong Wenchao, Principal Investigator, Universiti Putra Malaysia
Organization: Universiti Putra Malaysia (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024Y004
Record Dates: First submitted 2024-06-03; First posted 2024-06-21 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Physical Dependence
Keywords: Optimal load strength training;; neuromuscular adaptation;; long jumper; power output

STUDY DESIGN:
Intervention Model Description: In this study, the experimental group performed optimal load strength training aimed at developing the maximum power output of long jumpers, while the control group performed traditional strength training aimed at developing the fast strength of long jumpers.
Who Masked: Participant
Masking Description: Assistant coaches implementing the intervention plan.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group：power output (Experimental): by identifying the optimal load at which the athlete achieves the highest power output. The training program is then tailored based on these measurements, ensuring that the athlete trains at the load that maximizes their power output. This approach allows for more efficient and effective strength training, potentially leading to improved athletic performance. Throughout the training period, the VBT equipment continuously monitors the athlete's performance, providing real-time feedback and allowing for adjustments to the load as the athlete's strength and power improve. The goal is to enhance neuromuscular adaptations and optimize the athlete's power development, particularly during explosive movements like the vertical jump and long jump.
  Interventions: Other: Lower limb power output training
- Control Group:speed combined force (Experimental): Speed combined with strength training is designed to enhance the explosive power of long jumpers' lower limbs. This involves using maximum strength barbell squats and knee jumps to develop athletes' maximum strength and improve the speed of their neural contractions. Additionally, plyometric exercises and sprint drills are incorporated to further boost explosive power and coordination. This comprehensive training approach aims to optimize both the force and velocity aspects of power, leading to better overall performance in explosive movements critical for long jump success. Regular assessments and adjustments ensure that training loads are appropriate and effective for each athlete's progress.
  Interventions: Other: Force Combined Speed training

INTERVENTIONS:
Other: Lower limb power output training — Lower limb power output training content:
  Half squat up squat: 70%1R (6 repetitions × 5sets) + 5 knees jumps × 5 sets with an interval of 90 seconds；
  Arms: Experimental Group：power output
Other: Force Combined Speed training — Lower limb Force Combined Speed training content:
  Rapid half squat : Optimal load (6 sets × 7 repetitions). Rest intervals between sets range from 2 to 5 minutes.
  Arms: Control Group:speed combined force

SUMMARY:
The purpose of this study is to investigate the effects of optimal load strength training on the lower limb neuromuscular adaptation of athletes. An anatomical analysis of the vertical jump reveals three phases: the propulsion phase, the flight phase, and the landing phase.

This study is an 8-week randomized controlled trial. After selecting the participants, basic information such as height, weight, age, and years of training experience is collected. Subsequently, a maximal output power test for lower limb squatting is conducted. Participants are then randomly assigned to the speed group, power group, and strength group. The optimal power load for the power group is determined based on the participant maximal output power. Training plans are developed for the traditional group, power group, and strength group. Each training session is organized and supervised by a designated person. Surface electromyography, three-dimensional motion capture systems, and force platforms are used to collect electromyographic and kinetic data of participants during pre-test and post-test vertical jump actions. Electromyography evoked potential instruments and myotonometer are used to collect nerve signals of the tibial nerve (posterior calf) and muscle fiber dimension data of the rectus femoris before and after the experiment. Additionally, static full-range-of-motion vertical jump kinematics and kinetics data are collected before and after the experiment. To ensure the quality and validity of the intervention, the following controls are implemented during the experiment: first, communication with the participants to inform them of the purpose of the study and ensure adherence to the correct movement standards during testing; second, having a designated person responsible for resistance training during the experiment; third, using the same equipment and team for testing to maximize the controllability of the experiment process; fourth, providing verbal encouragement to participants during testing to maximize effort and minimize experimental errors. The aim is to determine the effects of optimal load strength training on improving the lower limb output power during the propulsion phase of the take-off stage in long jump athletes and the underlying neuromuscular adaptation mechanisms.

DETAILED DESCRIPTION:
In this study, the experimental group conducted 8 weeks of maximum output power strength training, and the control group also conducted 8 weeks of explosive power training (strength combined with speed). The subjects trained twice a week, and each training was not based on time, but on the number of times multiplied by the number of groups. The training load in the 8-week strength training of the experimental group was the load weight corresponding to the maximum output power of the subjects, and the training load in the control group was between 70% and 85% of the maximum strength. In the control group, the entire cycle was divided into three stages, 1-2 weeks: Adaptation period; 3-5 weeks: Enhancement period; 6-8 weeks: Stabilization period; the experimental group had no period division. The equipment for strength training in both the experimental and control groups was the Smith rack. The experimental group used weighted half squat jumps, and the control group used weighted half squat jumps plus knee hug jumps.

ELIGIBILITY:
Inclusion Criteria:

1. Aim for uniformity in various indicators to minimize errors caused by height, weight, and training experience differences.
2. Aim for a 1RM/body weight ratio of around 2.
3. Maintain normal diet and sleep patterns during the training period, and refrain from using supplements such as creatine and protein powder.
4. Male university long jump athletes should be aged ≥18, and they should not have engaged in strength training 48 hours before the baseline testing.

Exclusion Criteria:

1. Participants with various visceral diseases and abnormal liver or kidney function are excluded.
2. Those with unhealthy habits are excluded.
3. Participants with caffeine intake within 3 hours before testing are excluded.
4. Individuals who have engaged in high-intensity resistance exercises within the past 24 hours are excluded.
5. Those with lower limb joint injuries (open and closed) in the last 3 months are excluded.
6. Participants with contraindications such as cardiovascular diseases, skin allergies, and hernia are excluded.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Indicators of Neurological Adaptation（Number of nerve impulses） | From enrollment to the end of treatment at 8 weeks
  This includes the number of nerve impulses. Using wireless electromyography signal collection system
Muscle adaptation indicators (Muscle cross-sectional area) | From enrollment to the end of treatment at 8 weeks
  Muscle cross-sectional area assessment uses ultrasound to measure the cross-sectional area of the rectus femoris muscle fibers to assess muscle adaptation
Sports performance indicators (Vertical jump speed ) | From enrollment to the end of treatment at 8 weeks
  This study used three-dimensional motion capture equipment and a test bench to test the vertical jump speed of athletes.
Sports performance indicators (Power output) | From enrollment to the end of treatment at 8 weeks
  This study used three-dimensional motion capture equipment and a test bench to test the power output of athletes' lower limbs.
Sports performance indicators (Take-off height) | From enrollment to the end of treatment at 8 weeks
  This study used three-dimensional motion capture equipment and a test bench to test the athletes' take-off height before and after the experiment.
Indicators of Neurological Adaptation ( Nerve impulse frequency) | From enrollment to the end of treatment at 8 weeks
  This includes nerve impulse frequency，Using wireless electromyography signal collection system
Indicators of Neurological Adaptation (M wave amplitude) | From enrollment to the end of treatment at 8 weeks
  This includes the M wave amplitude，The test was performed using a potential evoked instrument.
Indicators of Neurological Adaptation (H-max/ M-max) | From enrollment to the end of treatment at 8 weeks
  This includes the H-max/ M-max. The test was performed using a potential evoked instrument. Among them, M-max refers to the average value of the first ten M-wave amplitude peaks. H-max refers to the maximum value of the H wave observed when the sensory nerve is stimulated at a frequency of 1Hz.
Indicators of Neurological Adaptation （Nerve conduction velocity） | From enrollment to the end of treatment at 8 weeks
  Nerve conduction velocity. The test was performed using a potential evoked instrument.
Indicators of Neurological Adaptation （Latency of the H reflex） | From enrollment to the end of treatment at 8 weeks
  Latency of the H reflex. The test was performed using a potential evoked instrument.
Indicators of Neurological Adaptation （presynaptic inhibition） | From enrollment to the end of treatment at 8 weeks
  This includes presynaptic inhibition. This value can only be obtained by processing the H reflex amplitude and the M wave amplitude. The presynaptic inhibition calculation formula is: Hmax1Hz = (Ave. H1:H10) / H1 PSI = Hmax1Hz / Mmax.

CONTACTS AND LOCATIONS:
Overall Officials: wenchao rong, Ph.D, Principal Investigator — University Putra Malaysia
Locations (2):
- China (2):
  - YanShan university, Qinhuangdao, HeiBei
  - Rong Wenchao, Qinhuangdao, HeiBei

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Sabido R, Hernandez-Davo JL, Botella J, Moya M. Effects of 4-Week Training Intervention with Unknown Loads on Power Output Performance and Throwing Velocity in Junior Team Handball Players. PLoS One. 2016 Jun 16;11(6):e0157648. doi: 10.1371/journal.pone.0157648. eCollection 2016. PMID 27310598
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/12872318/